CLINICAL TRIAL: NCT06174181
Title: Preventive TREatment of Dry Eye in Patients Receiving Repeated Intravitreal Injections for Age-related Macular Degeneration
Acronym: TREDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022PPRC11; 2023-A00620-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye Syndromes; Age-Related Macular Degeneration
MeSH Terms: conditions — Dry Eye Syndromes; Macular Degeneration

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Preservative-free ophtalmic lubricant emulsion countinuous during 6 month after intravitreal Injections for Age-related macular degeneration
  Interventions: Device: Preservative-free ophtalmic lubricant emulsion
- Routine treatment (Other): Preservative-free ophtalmic lubricant emulsion during few days after intravitreal Injections for Age-related macular degeneration
  Interventions: Other: Routine treatment

INTERVENTIONS:
Device: Preservative-free ophtalmic lubricant emulsion — Use of a preservative-free ophtalmic lubricant emulsion continous during 6 months
  Arms: Experimental
Other: Routine treatment — Use of a preservative-free ophtalmic lubricant emulsion after each intravitreal injection during few days
  Arms: Routine treatment

SUMMARY:
Age-related macular degeneration (AMD) is the 1st cause of visual impairment after the age of 50. Its most aggressive form, wet AMD, requires regular intravitreal injections (IVI) spaced 4 to 8 weeks apart usually depending on the treatment regimen and the patient's response. The IVI procedure requires a double disinfection with periocular and conjunctival cutaneous povidone-iodine. Antiseptic agents such as povidone iodine are a highly likely factor in the development of dry eye syndrome. Clinical data have demonstrated the abrasive and toxic effects of their use on the ocular surface, especially with repeated exposure (Saedon H, Nosek J, Phillips J. Ocular surface effects of repeated application of povisoden-iodine in patients receiving frequent intravitreal injections. Cutaneous and Ocular Toxicology. 2017;36(4):343-6.). The IVIS study coordinated by Prof. Dot reported impaired ocular surface and quality of life immediately after IVI. The authors suggest 3 levels of action to improve immediate tolerance: (i) improve the basal status of the ocular surface, (ii) reduce the contact time with povidone-iodine which could be toxic to the ocular surface and (iii) improve immediate post-IVI treatment. (Verrecchia S et al. A prospective multicentre study of intravitreal injections and ocular surface in 219 patients: IVIS study. Acta Ophthalmol. 2021 Mar 18). This study is part of the extension of the IVIS study. IVIs are effective and do not currently present a therapeutic alternative. However, their role in the development or exacerbation of dry eye is still poorly evaluated although millions of IVIs are performed each year worldwide (1.3 million in France in 2019). In addition, discomfort after injection is one of the factors that limit adherence to long-term IVI treatment, some patients fearing this repeated act. We propose in this bicentric, prospective, randomized, parallel group study, to evaluate in this context the impact of the continuous consideration of the risk of dry eye. The expected results are the objective improvement of dry eye indicators, comfort and quality of life of patients, all aimed at optimizing the adherence of our patients to their AMD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient treated for exudative AMD with at least one eye receiving IVI with an anti-VEGF for at least 12 months.
* Patient with at least one untreated dry eye symptom.
* Only one eye is included per patient. For patients injected bilaterally, the eye with the lowest TBUT will be included, otherwise the one with the highest Oxford score, otherwise the one with the lowest Schirmer score. If these 3 parameters are similar, the right eye will be included by default.
* Patient who has given informed consent to participate and understands the information related to the study.
* Patient affiliated with a social security plan or beneficiary of such a plan.
* Concurrent participation in non-interventional research is allowed. Concurrent participation in interventional research may be evaluated on a case-by-case basis by the Principal Investigator.

Exclusion Criteria:

* Patients with meatus plugs at inclusion.
* Eye surgery ≤ 3 months pre-inclusion (including laser or refractive).
* Anticholinergic* treatment prior to inclusion.
* Patients unable to maintain follow-up during the study period.
* Evidence of active ocular infection in either eye.
* History or presence of non-drying ocular surface disorders in either eye.
* Trauma or surgery to the eyelids.
* Any ocular or systemic pathology or treatment identified by the Investigator as likely to interfere with the results of the study.
* Hypersensitivity to any component of the medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Mean tear break-up time (TBUT) at the end of the study | 24 weeks
  Mean tear break-up time (TBUT) in seconds at the last study assessment. This is the standard measurement performed in routine care, which reduces the probability of missing data

SECONDARY OUTCOMES:
ocular surface alteration after 24 weeks | 24 weeks
  Ocular Staining Score d'Oxford

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Avicenne, Bobigny
  - HIA Desgenettes, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torres-Villaros H, Giocanti-Auregan A, Doan S, Agard E, Billant J, Arbousoff N, Matagrin B, Fenniri I, Dot C. Continuous versus Intermittent Use of Tear Substitutes in Patients Treated with Anti-VEGF for Neovascular Age-Related Macular Degeneration: The TREDIA Study. Ophthalmol Ther. 2025 Sep;14(9):2231-2241. doi: 10.1007/s40123-025-01201-3. Epub 2025 Jul 22. PMID 40691408